CLINICAL TRIAL: NCT05168501
Title: Assessing Variability of the Ventilatory Response to Duffin's Rebreathing Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Food and Drug Administration (FDA) (U.S. Federal Agency)
Collaborators: Spaulding Clinical Research LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SCR-013
Record Dates: First submitted 2021-12-13; First posted 2021-12-23 (Actual); Results first posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2021-12

CONDITIONS: Ventilation; Reproducibility; Physiology
Keywords: Duffin's rebreathing procedure; Ventilation; Pupillometry; Physiology
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: This study is an unblinded reproducibility assessment to assess variability of the ventilatory response to Duffin's rebreathing procedure. The lead-in reproducibility assessment will have up to 10 healthy volunteer participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lead-In (Experimental): Multiple rebreathing procedures using methodology developed by Duffin (referred to as Duffin's rebreathing procedure) will be conducted under hyperoxic and hypoxic conditions over the course of a day to confirm feasibility and gather reproducibility data using the procedure.
  Interventions: Other: Rebreathing procedure

INTERVENTIONS:
Other: Rebreathing procedure — Paired Duffin's rebreathing procedures performed two different isoxic end tidal PO2 levels (i.e., hyperoxic and hypoxic conditions) will be performed on Day 1 at 0, 2, 4, 6, and 24 hours.

SUMMARY:
This study will combine Duffin's rebreathing procedure with additional study procedures, such as quantitative pupillometry, that are planned for subsequent clinical studies in order to confirm feasibility and gather reproducibility data using the procedure. The reproducibility of Duffin rebreathing has been assessed previously by Mahamed and Duffin (2001) performing hyperoxic and hypoxic rebreathing procedures measured once daily for 14 consecutive days and then by Jensen et al. (2010) performing 4 pairs of hyperoxic and hypoxic rebreathing procedures in 1 day followed by 1 pair on 4 additional days separated by weeks to more than a month.

The present study is an unblinded reproducibility assessment to assess variability of the ventilatory response to Duffin's rebreathing procedure. Subjects will report to the study site for screening between Days -28 to -2 and then will return to the site on Day -1 for baseline assessments and check-in. After check-in (Day -1), subjects will remain in study site for PD assessments on Day 1 and check out on Day 2.

Paired rebreathing procedures (i.e., at two different isoxic end tidal PO2 [partial pressure oxygen] levels) will be performed on Day 1 at 0, 2, 4, and 6 hours. An additional pair of rebreathing procedures will be performed on Day 2 before checkout (approximately 24 hours). Subjects will not be administered any drugs in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject signs an Institutional Review Board (IRB)-approved written informed consent and privacy language as per national regulations (e.g., Health Insurance Portability and Accountability Act authorization) before any study related procedures are performed.
2. Subject is a healthy, non-smoking man or woman, 18 to 50 years of age, inclusive, who has a body mass index of 18.5 to 32 kg/m2, inclusive, at Screening.
3. Subject has normal medical history findings, clinical laboratory results, vital sign measurements, 12 lead ECG results, and physical examination findings at screening or, if abnormal, the abnormality is not considered clinically significant (as determined and documented by the investigator or designee).
4. Subject must have a negative test result for alcohol and drugs of abuse at screening and Check-in (Day -1).
5. Subject must test negative for severe acute respiratory syndrome coronavirus (SARS-CoV-2) by a molecular diagnostic test at check-in (Day -1). If a subject's test comes back inconclusive, it can be repeated at Check-in.
6. Female subjects must be of non-childbearing potential or, if they are of childbearing potential, they must: 1) have been strictly abstinent for 1 month before Check in (Day -1) and agree to remain strictly abstinent for the duration of the study and for at least 1-month after the last rebreathing procedure; OR 2) be practicing 2 highly effective methods of birth control (as determined by the investigator or designee; one of the methods must be a barrier technique) from at least 1 month before Check in (Day -1) until at least 1 month after the end of the study.
7. Male subjects must agree to practice 2 highly effective methods of birth control (as determined by the investigator or designee) from at least 1 month before Check In (Day -1) until at least 1 month after the last rebreathing procedure.
8. Subject is highly likely (as determined by the investigator) to comply with the protocol defined procedures and to complete the study.

Exclusion Criteria:

1. Subject has non-reactive or misshapen pupil(s) or damaged orbit structure or surrounding soft tissue is edematous or has an open lesion.
2. Subject Duffin rebreathing data is of poor quality or subject does not agree to remain clean-shaven for all days when the Duffin rebreathing procedure is being performed.
3. Subject has used any prescription or nonprescription drugs (including aspirin or NSAIDs and excluding oral contraceptives and acetaminophen) within 14 days or 5 half-lives (whichever is longer) or complementary and alternative medicines within 28 days before check-in.
4. Subject has used nicotine-containing products (e.g., cigarettes, cigars, chewing tobacco, snuff) within 6 weeks of Screening
5. Subject has a history or evidence of a clinically significant disorder, condition, or disease (e.g., cancer, human immunodeficiency virus [HIV], hepatic or renal impairment) that, in the opinion of the investigator would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion. This includes subjects with any underlying medical conditions that the Investigator believes would put subjects at increased risk of severe illness from COVID-19 based on the Centers for Disease Control and Prevention (CDC) guidelines.
6. Subject has any signs or symptoms that are consistent with COVID-19. These include subjects with fever or chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting, or diarrhea may have COVID-19. In addition, the subject has any other findings suggestive of COVID-19 risk in the opinion of the investigator.
7. Subject tests positive for SARS-CoV-2 by a molecular diagnostic test performed prior to admission.
8. Subject has clinical laboratory test results (hematology, serum chemistry and urinalysis) at Screening or Check-In that are outside the reference ranges provided by the clinical laboratory and considered clinically significant by the investigator.
9. Subject has a positive test result at Screening for HIV 1 or 2 antibody, hepatitis C virus antibodies, or hepatitis B surface antigen.
10. Female subject is pregnant or lactating before enrollment in the study.
11. Subject has a history of or currently has hypoventilation syndrome, sleep apnea, or chronic obstructive pulmonary disease (COPD) and is on non-invasive ventilation.
12. Subject has a history of asthma that has required medication within the last five years.
13. Subject has a history of sleep disorders, Panic Disorder, Panic Attacks, Generalized Anxiety Disorder, or any associated DSM diagnosis or condition.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2021-12-27 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Matousek, D.O., Principal Investigator — Spaulding Clinical Research LLC
Locations (1):
- Spaulding Clinical Research, West Bend, Wisconsin, United States

REFERENCES:
- [Background] Duffin J. Measuring the respiratory chemoreflexes in humans. Respir Physiol Neurobiol. 2011 Jul 31;177(2):71-9. doi: 10.1016/j.resp.2011.04.009. Epub 2011 Apr 14. PMID 21514404
- [Background] Mahamed S, Duffin J. Repeated hypoxic exposures change respiratory chemoreflex control in humans. J Physiol. 2001 Jul 15;534(Pt. 2):595-603. doi: 10.1111/j.1469-7793.2001.00595.x. PMID 11454975
- [Background] Jensen D, Mask G, Tschakovsky ME. Variability of the ventilatory response to Duffin's modified hyperoxic and hypoxic rebreathing procedure in healthy awake humans. Respir Physiol Neurobiol. 2010 Feb 28;170(2):185-97. doi: 10.1016/j.resp.2009.12.007. Epub 2009 Dec 24. PMID 20035904

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was halted after 7 participants as sufficient experience with the experimental technique was obtained to move on to subsequent studies.
Period: Overall Study
Arm/Group | Lead-In
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lead-In
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.6 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Baseline Minute Ventilation
Description: Minute ventilation during the rebreathing assessment when end tidal PCO2 (partial pressure carbon dioxide) is less than the ventilatory recruitment threshold (represents non-chemoreflex drives to breathe; 'flat' portion of minute ventilation versus end tidal PCO2 relationship). Data was analyzed using linear-mixed effects regression of baseline minute ventilation with random effects for between subject, between day, and between occasion variability. Reported value is the mean for the treatment group across all individuals, days, and times.
Time Frame: 0, 2, 4, 6 and 24 hours
Population: All participants who successfully completed one rebreathing assessment.
Measure: Mean (Standard Deviation); unit: L/min
Groups:
- Hyperoxic Rebreathing: Multiple rebreathing procedures using methodology developed by Duffin (referred to as Duffin's rebreathing procedure) were conducted under hyperoxic conditions (maintained isoxic 150 mmHg) at 0, 2, 4, 6, and 24 hours.
- Hypoxic Rebreathing: Multiple rebreathing procedures using methodology developed by Duffin (referred to as Duffin's rebreathing procedure) were conducted under hypoxic conditions (maintained isoxic 50 mmHg) at 0, 2, 4, 6, and 24 hours.
Arm/Group | Hyperoxic Rebreathing | Hypoxic Rebreathing
Number analyzed (Participants) | 7 | 7
L/min | 11.6 (3.4) | 12.0 (2.9)

2. Primary Outcome: Ventilatory Recruitment Threshold
Description: The end tidal PCO2 point above which minute ventilation starts to increase linearly with further increases in end tidal PCO2. Data was analyzed using linear-mixed effects regression of ventilatory recruitment threshold with random effects for between subject, between day, and between occasion variability. Reported value is the mean for the treatment group across all individuals, days, and times.
Time Frame: 0, 2, 4, 6 and 24 hours
Population: All participants who successfully completed one rebreathing assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Hyperoxic Rebreathing | Hypoxic Rebreathing
Number analyzed (Participants) | 7 | 7
mmHg | 43.0 (3.0) | 38.1 (1.7)

3. Primary Outcome: Slope of the PCO2-ventilatory Response Curve
Description: Slope of the minute ventilation versus end tidal PCO2 curve that reflects the increase in minute ventilation relative to the increase in end tidal PCO2. Data was analyzed using linear-mixed effects regression of Slope of the PCO2-ventilatory response curve with random effects for between subject, between day, and between occasion variability. Reported value is the mean for the treatment group across all individuals, days, and times.
Time Frame: 0, 2, 4, 6 and 24 hours
Population: All participants who successfully completed one rebreathing assessment.
Measure: Mean (Standard Deviation); unit: L/min/mmHg
Arm/Group | Hyperoxic Rebreathing | Hypoxic Rebreathing
Number analyzed (Participants) | 7 | 7
L/min/mmHg | 3.19 (2.46) | 3.28 (2.41)

4. Primary Outcome: Extrapolated Ventilatory Recruitment Threshold
Description: Intersection of the slope of the PCO2-ventilation response curve with the X axis. Data was analyzed using linear-mixed effects regression of extrapolated ventilatory recruitment threshold with random effects for between subject, between day, and between occasion variability. Reported value is the mean for the treatment group across all individuals, days, and times.
Time Frame: 0, 2, 4, 6 and 24 hours
Population: All participants who successfully completed one rebreathing assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Hyperoxic Rebreathing | Hypoxic Rebreathing
Number analyzed (Participants) | 7 | 7
mmHg | 36.8 (7.1) | 32.7 (5.9)

ADVERSE EVENTS:
Time Frame: 2 days
Groups:
- Hyperoxic Rebreathing: Multiple rebreathing procedures using methodology developed by Duffin (referred to as Duffin's rebreathing procedure) will be conducted under hyperoxic conditions (maintained isoxic 150 mmHg) at 0, 2, 4,6, and 24 hours.
Arm/Group | Hyperoxic Rebreathing | Hypoxic Rebreathing
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-09): https://cdn.clinicaltrials.gov/large-docs/01/NCT05168501/Prot_SAP_000.pdf